CLINICAL TRIAL: NCT05937763
Title: Feasibility and Evaluation of an Adaptive STaffing Model in a Community Emergency Department (FAST-ED)
Brief Title: ED Adaptive Staffing Study
Acronym: FAST-ED
Status: Recruiting | Type: Observational
Sponsor: Oak Valley Health (Other)
Responsible Party: Sponsor
Other Study IDs: 148-2306
Record Dates: First submitted 2023-06-23; First posted 2023-07-10 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Emergency Medicine; Well-Being, Psychological
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Primary Care Paramedic (PCP) Block: A PCP will be staffed in the emergency department offload zone 3 days a week (Monday, Wednesday, and Friday) on a 10am - 10pm shift, in addition to the standard staffing model.
  Interventions: Other: Staffing model
- Registered Nurse (RN) Block: An experienced emergency department RN with triage training will be staffed in the emergency department offload zone 3 days a week (Monday, Wednesday, and Friday) in a 10am - 10pm shift, in addition to the standard staffing model
  Interventions: Other: Staffing model
- Current Workflow Block: The currently hospitals staffing models of the emergency department offload zone.

INTERVENTIONS:
Other: Staffing model — Staffing the hospitals emergency department offload zone with a PCP or RN or current workflow.
  Groups: Primary Care Paramedic (PCP) Block; Registered Nurse (RN) Block

SUMMARY:
Emergency Departments (EDs) across Ontario are being inundated with unprecedented high patient volumes and a staffing shortage that directly impacts patient care and flow. An area of concern among EDs is the offload zone where patients are brought in by ambulance. EMS offload time is the time it takes paramedics to transfer a patient to the appropriate area within an emergency department and give hospital staff a summary of what concerns the patient is seeking care for. There are multiple factors that may delay this time, including limited staff in the offload area to complete the transfer process due to competing patient care responsibilities. The adaptive staffing model study will look to add a primary care paramedic (PCP) or a registered nurse (RN) in the offload zone during times of high ambulance volume (August to January) to help with patient care within the offload zone. This single-centered community hospital study will evaluate the benefits of having a PCP or RN, compared to the current model, on ambulance offload times, patient safety outcomes, patient treatment times, and staff well-being using three different models of staffing.

ELIGIBILITY:
Inclusion Criteria:

* Patients brought in by ambulance to hospitals emergency department offload area

Exclusion Criteria:

* Patients not arriving to the hospitals emergency department offload area

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will use a convenience sampling method, given that patients brought in by ambulance are at random and non-predictive.
Sampling Method: Non-Probability Sample
Enrollment: 5917 (Estimated)
Dates: Start 2023-10-02 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Triage Time | 6 months
  The aim of this objective is to compare time to triage and time to transfer of care for three models of staffing.
Return to Service | 6 months
  The aim of this objective is to determine if an adaptive staffing model during peak volumes reduces ambulance offload times and return to service.

SECONDARY OUTCOMES:
Time to provider assessment | 6 months
Provider Feedback Survey | 6 months
  Explore provider perceptions (ED staff and paramedics) of each model with the aim of determining which model provides better patient care during peak volumes. Participants will self-report their perceived barriers, challenges and benefits of the staffing interventions.
Time to treatment | 6 months
Time to disposition | 6 months
Number of incident reports | 6 months
  Patient safety events
Case costing | 6 months
Well-being Index (questionnaire) | 6 months
  Explore staff and paramedic well-being on intervention model

CONTACTS AND LOCATIONS:
Locations (1):
- Markham Stouffville Hospital, Markham, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Aggregate data and study results will be shared via publication and conference presentations.